CLINICAL TRIAL: NCT05913804
Title: An Exploratory Clinical Study on the Safety and Efficacy of YTS104 Cell Injection in the Treatment of Relapsed or Refractory Multiple Myeloma
Brief Title: YTS104 Cell Injection for the Treatment of Relapsed or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023020
Record Dates: First submitted 2023-05-11; First posted 2023-06-22 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-09

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- YTS104 cells injection (Experimental): Subjects will receive cell infusion, with the initial cell dose of 1E6/kg. 1-6 subjects will be enrolled. The second dose group was 3E6 cells /kg with 1-6 subjects; The third and fourth dose groups were 6E6 cells /kg and 1E7 cells /kg, respectively, with 3-6 subjects.Subjects may undergo secondary or multiple retransfusion
  Interventions: Biological: YTS104 Cells injection

INTERVENTIONS:
Biological: YTS104 Cells injection — YTS104 Cell injection(LILRB4 dual STAR-T Cell Injection/BCMA LILRB4 Dual STAR-T Cell Injection)) is a new STAR-T cell transfected by lentivirus.The study required that lymphocytes were collected from the subjects and cultured for 2-3 weeks to obtain YTS104 cell injection. Subjects were treated with fludarabine and cyclophosphamide chemotherapy prior to reinfusion, followed by a 2-day rest period before cell infusion.

SUMMARY:
This is a single-center, single-arm, open-label phase I clinical study to determine the safety and efficacy of relapsed or refractory multiple myeloma subjects

DETAILED DESCRIPTION:
This study will recruit multiple myeloma subjects,and Subjects should undergo FC chemotherapy before returning the cells, then followed by infusion of YTS104 cells injection. YTS104 cells injection will be intravenously infused with a escalated dose of 1E6#3E6#6E6#1E7 cells/kg.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years, gender is not limited;
* Patients diagnosed as relapsed/refractory multiple myeloma according to the International Myeloma Working Group (IMWG 2014) criteria for multiple myeloma after at least 3 lines of treatment (including at least one proteasome inhibitor and an immunomodulator based chemotherapy regimen), and at least one complete treatment cycle per line of treatment; Documented disease progression during or within 12 months after the most recent antimyeloma therapy (not limited to 12 months after CAR-T therapy as the last line of therapy);
* The presence of one or more measurable lesions at screening was defined as any of the following: 1) serum M-protein ≥0.5g/dL (≥5g/L), 2) urinary M-protein level ≥200 mg/24 hours; 3) serum free light chain (sFLC) ≥100 mg/L and serum κ/λ free light chain ratio abnormal (<0.26 or >1.65);
* Good organ function;
* ECOG score ≤1;
* The predicted survival time was ≥12 weeks;
* Female subjects of childbearing age or male subjects with partners of women of childbearing age agreed to use effective methods of contraception throughout the trial and for 12 months after cell infusion;
* The subjects voluntarily participated in the study, signed the informed consent form, and complied with the follow-up.

Exclusion Criteria:

* A history of allergy to any component of the cell product;
* Patients who had used CAR-T cell therapy or any other gene transduction or other therapeutic products within 3 months after signing the informed consent, except those with undetectable CAR-T cells or CAR-T cells below the lower limit of detection;
* Subjects had plasma cell leukemia, Waldenström's macroglobulinaemia, POEMS syndrome, or primary light chain amyloidosis;
* Patients with a history of any of the following cardiovascular and cerebrovascular diseases within the preceding 6 months were screened;

  1. Congestive heart failure (New York Heart Association [NYHA]≥III), congenital long QT syndrome, left front half block (double bundle block), asymptomatic right bundle branch block allowed; Myocardial infarction, unstable angina pectoris, coronary angioplasty, stent implantation, coronary/peripheral artery bypass grafting;
  2. Cerebrovascular accident (CVA) and transient ischemic attack (TIA);
  3. Severe arrhythmias requiring treatment (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes, etc.); d: Subjects had uncontrolled hypertension (systolic blood pressure greater than 160 mmHg and/or diastolic blood pressure greater than 100 mmHg), a history of hypertensive crisis, or hypertensive encephalopathy;
* Pulmonary embolism, or deep venous thrombosis of the lower extremity requiring anticoagulation, or active lung disease and/or pneumonia have occurred within 6 months prior to screening;
* Hepatitis B surface antigen (HBsAg) positive; Hepatitis B core antibody (HBcAb) and HBV DNA in peripheral blood were positive. Hepatitis C virus (HCV) antibody positive and HCV RNA positive; Treponema pallidum antibody was positive;
* Patients with known systemic lupus erythematosus, co-active or uncontrolled autoimmune diseases (e.g., Crohns disease, rheumatoid arthritis, autoimmune hemolytic anemia, etc.), primary or secondary immunodeficiency (e.g., HIV infection or severe infectious diseases);
* Patients with previous or concurrent uncured malignant tumors with unstable control, affecting the long-term survival of the subjects, excluding cured cervical carcinoma in situ, non-invasive basal cell or squamous cell skin cancer, or other malignant tumors with local prostate cancer after radical treatment, ductal carcinoma in situ after radical treatment and no recurrence for at least 5 years;
* Patients with current or previous history of central nervous system disease, such as seizures, stroke, severe brain injury, aphasia, paralysis, dementia, Parkinson's disease, mental illness, etc.;
* Have central nervous system (CNS) involvement or symptoms of CNS involvement (including cranial neuropathy and extensive lesions or spinal cord compression);
* Patients had undergone previous solid-organ transplantation or allogeneic hematopoietic stem-cell transplantation (allo-HSCT) 6 months before screening or autologous stem-cell transplantation within 3 months before apheresis;
* Patients with acute or chronic graft-versus-host disease (GVHD) at screening time;
* The following anti-MM treatments were used at the indicated times prior to apheresis:

  1. Use of any immunosuppressant or radiotherapy within 2 weeks prior to apheresis;
  2. Received cytotoxic or proteasome inhibitors or small-molecule targeted therapy within 2 weeks of preapheresis or 3 half-lives, whichever is shorter;
  3. Received any macromolecular therapy such as monoclonal antibodies within 4 weeks prior to anapheresis or within 3 half-lives, whichever is shorter;
  4. Received immunomodulator within 1 week;
* The patient had a history of live vaccination within 4 weeks before signing ICF;
* Subjects had a history of mental illness, or substance abuse;
* Subjects were pregnant or lactating;
* If participating in other interventional clinical studies before apheresis, the requirements of drug washout before apheresis should be met;
* The investigator believes that there are other factors unsuitable for inclusion or affecting participants' participation in or completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | Within 28 days after cell transfusion
  Dose-limiting toxicity was defined as adverse events associated with YTS104-cell injection within 28 days of cell transfusion, including grade 4 or 5 CRS and ICANS; grade 4 haematological adverse events did not return to grade 2 or baseline within 28 days of cell transfusion
Incidence and severity of adverse events | 24 months
  After YTS104-cell infusion, adverse events will be graded as CTCAE 5.0

SECONDARY OUTCOMES:
Overall response rate (ORR) | 24 months
  Including sCR, CR, VGPR, and PR.
Duration OF RESPONSE(DOR) | 24 months
  DOR was defined as the time from the first documentation of response (PR or better) to the first documentation of disease progression or death from any cause after YTS104 infusion in patients with PR or better.
Progression-free survival(PFS) | 24 months
  PFS was defined as the time between the subject's YTS104-cell infusion and the occurrence of disease progression or death from any cause.
Overall survival(OS) | 24 months
  It was defined as the time between the subject's reinfusion of YTS104 cell injection and death from any cause.
Expansion and persistence of YTS104 cell injection in vivo | 24 months
  The proportion of STAR-T in peripheral blood was detected by flow cytometry,The copies of STAR-T DNA in peripheral blood was detected by qPCR method.

CONTACTS AND LOCATIONS:
Overall Officials: Gang An, Study Director — Institute of Hematology & Blood Diseases Hospital Ethics Committee; Lugui Qiu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital Ethics Committee
Locations (1):
- Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No